CLINICAL TRIAL: NCT02014649
Title: Randomised, Parallel Dose, Phase 1/2 Safety and Pharmacokinetics Study of Inhaled Laninamivir Octanoate TwinCaps® Dry Powder Inhaler in Children With Naturally Acquired Influenza A or B
Brief Title: Safety & Pharmacokinetics Study of Inhaled Laninamivir Octanoate TwinCaps® Dry Powder Inhaler in Children With Influenza
Acronym: FROSTY
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Study was terminated as per BARDA decision to terminate contract.
Sponsor: Biota Scientific Management Pty Ltd (Industry)
Collaborators: Department of Health and Human Services (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: Vaxart (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: BTA51-350-203; U1111-1150-7392 (Other: WHO)
Record Dates: First submitted 2013-11-24; First posted 2013-12-18 (Estimated); Results first posted 2025-01-13 (Actual); Last update posted 2025-01-13 (Actual); Status verified 2025-01

CONDITIONS: Influenza
Keywords: Influenza treatment; pediatric; laninamivir
MeSH Terms: conditions — Influenza, Human | interventions — laninamivir; CS 8958; Lactose

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 20mg Laninamivir Octanoate (Experimental): Dry Powder plus placebo
  Interventions: Drug: 20 mg laninamivir octanoate; Drug: Placebo
- 40mg Laninamivir Octanoate (Experimental): Dry Powder
  Interventions: Drug: 40 mg laninamivir octanoate

INTERVENTIONS:
Drug: 20 mg laninamivir octanoate
  Other Names: CS-8958
  Arms: 20mg Laninamivir Octanoate
Drug: Placebo
  Other Names: Lactose
  Arms: 20mg Laninamivir Octanoate
Drug: 40 mg laninamivir octanoate
  Other Names: CS-8958
  Arms: 40mg Laninamivir Octanoate

SUMMARY:
This Phase 1/2 protocol is designed to collect safety, tolerability and pharmacokinetic data of two doses of Laninamivir Octanoate in children and adolescents. The protocol will also explore virology and efficacy endpoints.

DETAILED DESCRIPTION:
Approximately 48 subjects aged 5-17 years inclusive will be randomised into the study.

Subjects with recent onset of presumptive influenza will have influenza A or B infection confirm by Rapid Antigen Test.

The study will be conducted on an outpatient basis. The dose is administered in a single session in the clinic on Day 1. The subject will return to the clinic for assessments and follow up.

ELIGIBILITY:
Inclusion Criteria:

* Subjects' parent/legally acceptable representative/guardian must give written informed consent to participate in the study and must understand the nature of the study and must be willing to comply with all protocol requirements. Subjects over 12 must provide assent to participate in the study and potential subjects below this age should provide assent if deemed appropriate to the maturity level of the subject or if required according to local guidance/regulations.
* Males or females aged between 5 and 17 years inclusive, who weigh at least 15 kg at screening.
* Confirmed influenza infection based on positive rapid antigen test (RAT) for Influenza A or B.
* Fever, defined as either:

  1. Otic temperature ≥38.0° C (100.4°F) at the screening visit, OR,
  2. A history of fever within the 24 hours prior to the screening visit and has administered antipyretic(s) in the 6 hours prior to the screening visit.
* Presence on the Screening questionnaire of, at least two, of the following influenza symptoms:

  1. Non-productive Cough, of at least moderate severity,
  2. Sore throat, of at least moderate severity,
  3. Nasal congestion/runny nose, of at least moderate severity,
  4. Headache, of at least moderate severity,
  5. Muscle aches and pain, of at least moderate severity,
  6. Feeling feverish, of at least moderate severity,
  7. Low energy, tired, fatigue, of at least moderate severity;
* Onset of illness no more than 40 hours before randomization, defined as:

  1. time when the temperature was first measured as elevated ≥38.0°C (oral or otic) OR
  2. time when the subject first experienced at least one influenza symptom (non-productive cough, sore throat or nasal congestion/runny nose, headache, muscle aches and pain, feeling feverish, or low energy/tired/fatigue)
* In the Investigator's opinion able to complete the required inhalations of the investigational medicinal product.

Exclusion Criteria:

* Use of antiviral treatment for influenza (e.g., zanamivir, oseltamivir, peramivir, rimantadine, or amantadine) within 14 days prior to screening
* Received influenza virus vaccine in the previous 3 weeks.
* History or presence of clinically significant pulmonary disease (e.g., chronic obstructive pulmonary disease, cystic fibrosis, or bronchiectasis)
* Current asthma requiring treatment, or history of asthma requiring treatment in the last 5 years, or episode of wheezing in the 12 months prior to randomization.
* History of congestive heart failure with symptoms consistent with New York Heart Association Class III or IV functional status.
* Presence of an immune compromised status due to chronic illness, organ transplantation or use of daily systemic immunosuppressants
* Presence of clinically significant signs of acute respiratory distress during screening.
* Current use of inhaled medications (nasal or oral) or anticipated use of inhaled medications (nasal or oral) at any time during the study.
* Current or a history of acute or chronic renal impairment/disease
* Currently hospitalized or any planned hospitalizations within 1 month following the last dose of IMP.
* Current clinical evidence of otitis, bronchitis, sinusitis, or pneumonia or active bacterial infection at any body site
* Severe infection within 30 days prior to screening which required parenteral antibiotic use or hospitalization.

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 15 (Actual)
Dates: Start 2013-11; Primary Completion 2014-04 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jolanta Airey, Dr, Study Director — Biota Scientific Management Pty Ltd
Locations (28):
- United States (28):
  - Precision Trials LLC, Phoenix, Arizona
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - SoCal Clinical Research Med Group, Bellflower, California
  - Sherif Khamis MD Inc, Canoga Park, California
  - Advanced Medical Research, Lakewood, California
  - Madera Family Medical Group, Madera, California
  - Connecticut Children's Medical Center, Hartford, Connecticut
  - A.G.A Clinical Trials, Hialeah, Florida
  - Lafayette Clinical Research Group, Lafayette, Indiana
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - Louisiana State University Health Sciences Center, Shreveport, Louisiana
  - Dr Haidar's Clinic, Carriere, Mississippi
  - DePaul Health Center, Bridgeton, Missouri
  - Blue Ridge Pediatric and Adolescent Medicine Group, Boone, North Carolina
  - Dayton Children's Hospital, Dayton, Ohio
  - The University of Toledo Medical Center, Toledo, Ohio
  - Dr Santiago Reyes, Oklahoma City, Oklahoma
  - Cyn3rgy Research, Gresham, Oregon
  - Sanford Research University of South Dakota, Sioux Falls, South Dakota
  - Avant Research Assoc., Houston, Texas
  - West Houston Clinical Research Service, Houston, Texas
  - Foothill Family Clinic, Salt Lake City, Utah
  - First Med, Salt Lake City, Utah
  - Foothill Family Clinic South, Salt Lake City, Utah
  - Copperview Medical Center, South Jordan, Utah
  - Dixie Pediatrics, St. George, Utah
  - Rockwood Clinic, Spokane, Washington
  - Rockwood North Clinic, Spokane, Washington

RESULTS

PARTICIPANT FLOW:
Groups:
- 20mg Laninamivir Octanoate: Dry Powder plus placebo
  20 mg laninamivir octanoate
  Placebo
- 40mg Laninamivir Octanoate: Dry Powder
  40 mg laninamivir octanoate
Period: Overall Study
Arm/Group | 20mg Laninamivir Octanoate | 40mg Laninamivir Octanoate
Started | 7 | 8
Completed | 7 | 8
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 20mg Laninamivir Octanoate | 40mg Laninamivir Octanoate | Total
Number analyzed (Participants) | 7 | 8 | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 7 | 8 | 15
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 8.3 (3.77) | 9.8 (2.82) | 9.1 (3.26)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 4 | 8
  Male | 3 | 4 | 7
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 7 | 8 | 15

OUTCOME MEASURES:

1. Primary Outcome: To Evaluate Time to First Alleviation of a Composite of Influenza Symptoms and Absence of Fever.
Description: For subjects aged 5 through 12 years, the subject or parent/legal guardian completed the Canadian Acute Respiratory Illness and Flu Scale (CARIFS) symptom diary and measured otic body temperature twice a day, in the morning between 6 and 10AM and evening between 6 and 10PM, until the Day 10 visit. Subjects aged 13 through 17 years completed the Influenza Symptom Questionnaire (ISQ) themselves and measured otic body temperature twice a day, in the morning between 6 and 10AM and evening between 6 and 10PM, until the Day 10 visit.
Time Frame: Subjects are assessed at clinic visits and followed up to 28-days post dose.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | 20mg Laninamivir Octanoate | 40mg Laninamivir Octanoate
Number analyzed (Participants) | 6 | 8
hours | 85.1 (34.2) | 79.7 (29.8)

2. Secondary Outcome: To Evaluate the Pharmacokinetic (PK) Profiles (Concentration) of the Prodrug, Laninamivir Octanoate, and Its Active Metabolite, Laninamivir, Following Administration of a Single Dose (20 or 40 mg)
Description: Pharmacokinetic parameters will be calculated and summarized, PK concentration data will add to population models.
Time Frame: Samples are collected at clinic visits over 5 days.
Population: Due to early study termination, no PK data were collected.
Arm/Group | 20mg Laninamivir Octanoate | 40mg Laninamivir Octanoate
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | 20mg Laninamivir Octanoate | 40mg Laninamivir Octanoate
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/8
Other Adverse Events (participants affected / at risk) | 2/7 | 5/8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 20mg Laninamivir Octanoate (N=7) | 40mg Laninamivir Octanoate (N=8)
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Rhinitis Allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Otitis Media Bacterial (Infections and infestations) | 0 | 1
Tonsillitis Bacterial (Infections and infestations) | 1 | 0
Urinary Tract Infection (Infections and infestations) | 1 | 0
Skin Discolouration (Skin and subcutaneous tissue disorders) | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1
Tympanic Membrane Disorder (Ear and labyrinth disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 0 | 1

LIMITATIONS AND CAVEATS:
Sponsor's decision to terminate the study based on funding considerations and equivocal results from a Phase 2 study in adults (BTA51-350-201). As a result, the full prospectively planned efficacy analyses were not completed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes